CLINICAL TRIAL: NCT05280028
Title: The Impact of Different Hormone Therapy Regimens on Overactive Bladder Symptoms, Sexual Function, Depressive Symptoms, Autonomic Function, and Arterial Stiffness
Brief Title: HRT on Overactive Bladder Symptoms, Sexual Function, Depressive Symptoms, Autonomic Function, and Arterial Stiffness
Status: Recruiting | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief of Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 110262-F
Record Dates: First submitted 2022-02-23; First posted 2022-03-15 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Menopausal Syndrome
MeSH Terms: interventions — tibolone; Estradiol; Medroxyprogesterone Acetate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tibolone: Tibolone 2.5 mg per day
  Interventions: Drug: Tibolone 2.5 mg
- Indivina: Estradiol valerate (E2V) 1mg & medroxyprogesterone acetate 2.5 mg (MPA) per day
  Interventions: Drug: Estradiol valerate 1 mg/medroxyprogesterone acetate 2.5 mg

INTERVENTIONS:
Drug: Tibolone 2.5 mg — Tibolone 2.5 mg per day
  Other Names: Livial
  Groups: Tibolone
Drug: Estradiol valerate 1 mg/medroxyprogesterone acetate 2.5 mg — Estradiol valerate 1 mg/medroxyprogesterone acetate 2.5 mg per day
  Other Names: Indivina
  Groups: Indivina

SUMMARY:
Therefore, the aim of this study is to assess the therapeutic effect on overactive bladder symptoms, sexual function, heart rate variability, arterial stiffness, atherosclerosis, sleep, and depression between tibolone and E2V/MPA.

From the results, the investigators will compare the effect of tibolone versus E2V/MPA on overactive bladder symptoms, sexual function, autonomic function, arterial stiffness, atherosclerosis, sleep and depression.

DETAILED DESCRIPTION:
Menopausal syndromes include overactive bladder symptom, autonomic symptoms, and even sexual dysfunction. Hormone therapy (HT) is widely used for controlling menopausal symptoms. Common HT for menopausal syndrome with intact uterus includes tibolone, estradiol valerate (E2V) 1mg & medroxyprogesterone acetate (MPA), and conjugated equine estrogens (CEE) & MPA.

However, only a few literatures mentioned about the therapeutic effect of tibolone, but lack of comparison research about their therapeutic effect on overactive bladder symptoms, sexual function, heart rate variability, arterial stiffness, atherosclerosis, sleep and depression. The knowledge of the above therapeutic effects should be important for choosing a suitable medication. Therefore, the aim of this study is to assess the therapeutic effect on overactive bladder symptoms, sexual function, heart rate variability and arterial stiffness between tibolone and E2V/MPA.

All female patients with intact uterus who underwent treatment for menopausal syndrome at Far Eastern Memorial Hospital from October 2021 will be included. An open-labeled, prospective, comparative study design will be used. HT included tibolone (2.5 mg/day) or E2V (1mg) & MPA (2.5 mg) per day. The enrolled women will be requested to complete the Greene climacteric scale, Urgency Severity Scale, Overactive Bladder Symptom Score, the International Prostate Symptom Score (IPSS), the Female Sexual Function Index (FSFI), the Pittsburgh Sleep Quality Index, Center for Epidemiological Studies Depression questionnaire, heart rate variability, arterial stiffness and atherosclerosis examinations at baseline, and 4 weeks (visit 2) and 12 weeks (visit 3) after treatment.

From the results, the investigators will compare the effect of tibolone versus E2V/MPA on overactive bladder symptoms, sexual function, autonomic function, arterial stiffness, atherosclerosis, sleep and depression. Currently, there is no similar research as our current study.

ELIGIBILITY:
Inclusion Criteria:

* >20 years old female
* Menopausal symptoms, still have a uterus, and no breast or other cancers, and no vascular-blocking disease such as stroke.

Exclusion Criteria:

* Nil.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: Women with menopausal symptoms
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overactive bladder symptoms | 3 months
  Compare the effect of tibolone versus E2V/MPA on the total score of Overactive Bladder symptoms Score Total scores:0-15, the minimum values and whether lowest scores mean a better outcome
Sexual function index | 3 months
  Compare the effect of tibolone versus E2V/MPA on total score of the Female Sexual Function Index Total scores:4-95, the maximum values and whether higher scores mean a better outcome.
Autonomic function | 3 months
  Compare the effect of tibolone versus E2V/MPA on heart rate variability parameters
Arterial stiffness | 3 months
  Compare the effect of tibolone versus E2V/MPA on cardio-ankle vascular index

SECONDARY OUTCOMES:
Atherosclerosis | 3 months
  Compare the effect of tibolone versus E2V/MPA on ankle-brachial pressure index

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Mou Hsiao, MD, Principal Investigator — Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital
Locations (1):
- Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan